CLINICAL TRIAL: NCT05676476
Title: The ACHIEVE Trial: Achieving Longer Gestation in Preeclampsia Via Antihypertensive Therapy.
Acronym: Achieve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rachel Sinkey, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23HL159331 (NIH); 1K23HL159331 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia; Gestational Hypertension; Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Toxemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Antihypertensive treatment for a BP goal of less than 140/90 mmHg
  Interventions: Drug: Antihypertensive treatment
- Usual Care (No Intervention): Antihypertensive treatment only if BP ≥ 160/110 mmHg

INTERVENTIONS:
Drug: Antihypertensive treatment — Antihypertensive treatment to goal of less than 140/90 mmHg
  Arms: Intervention

SUMMARY:
The Achieve Trial is a randomized clinical trial to test whether lowering blood pressure to less than 140/90 mmHg in women with hypertensive disorders of pregnancy will prolong pregnancy.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy, including gestational hypertension and preeclampsia, are characterized by new onset high blood pressure in pregnancy and constitute a major cause of maternal and perinatal morbidity and mortality; severe hypertension (blood pressure ≥160/110 mmHg) is a common trigger for antihypertensive treatment and preterm delivery. We propose a clinical trial that will test whether lowering the blood pressure in women with hypertensive disorders of pregnancy at <36 weeks' gestation to <140/90 mmHg will prolong pregnancy and, therefore, improve maternal and fetal/neonatal outcomes. Data generated in this study, along with knowledge and skills acquired by the candidate in the complementary career development plan, will facilitate an independent research career focused on hypertension and cardiovascular disease in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Gestational age: 23 weeks, 0 days to 35 weeks, 6 days
* Hypertensive disorder of pregnancy including gestational hypertension or preeclampsia, the non-severe form at enrollment, which is called without severe features by the American College of Obstetricians and Gynecologists.
* No evidence of the severe form of preeclampsia, termed severe features, as outlined in maternal exclusions
* No indication for delivery at the time of enrollment.
* Planned expectant management at time of enrollment
* Singleton or dichorionic twin gestation, defined at and beyond 14 weeks gestation. (A pregnancy complicated by a vanishing twin in the first trimester defined as less than 14 weeks gestation will be eligible.)
* Intact membranes

Exclusion Criteria:

* Preeclampsia with severe features, defined per ACOG as:
* Systolic blood pressure of 160 mm Hg or more, or diastolic blood pressure of 110 mm Hg or more on two occasions at least 4 hours apart (unless antihypertensive therapy is initiated before this time)
* Thrombocytopenia defined as: lower than 100 x 10e9 platelets/L
* Impaired liver function that is not accounted for by alternative diagnoses and as indicated by abnormally elevated blood concentrations of liver enzymes (to more than twice the upper limit normal concentrations), or by severe persistent right upper quadrant or epigastric pain unresponsive to medications
* Renal insufficiency (serum creatinine concentration more than 1.1 mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease)
* Pulmonary edema
* New-onset headache unresponsive to medication and not accounted for by alternative diagnoses
* Visual disturbances
* Underlying renal dysfunction defined as, presenting the following parameters prior to 20 weeks gestation: baseline creatinine, equal to or higher than, 1.2 mg/dL Or proteinuria: defined as presenting protein in urine, equal to or higher than, 300 mg/24 hours or protein/creatinine ratio, equal to or higher than, 0.3 or Urine dipstick reading of greater than or equal to 2 at baseline and in the absence of a urinary tract infection
* Stage 2 chronic hypertension
* Contraindications to labetalol and nifedipine XL according to the FDA package insert
* Patient unable to or unwilling to adhere to management recommendations
* Fetal Reasons for Study Ineligibility:
* Fetal growth restriction (lower than 10th percentile) at enrollment, based on an ultrasound within 3 weeks prior to enrollment
* Oligohydramnios defined by amniotic fluid deepest vertical pocket <2 cm based on an ultrasound within the 48 hours prior to enrollment
* Known major structural or chromosomal abnormality

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean number of days from randomization to delivery | From randomization to delivery, up to 14 weeks
  Duration of prolongation of pregnancy

SECONDARY OUTCOMES:
Perinatal morbidity | 6 weeks
  Composite of NICU admission ≥2 days, bronchopulmonary dysplasia, necrotizing enterocolitis, intraventricular hemorrhage, retinopathy of prematurity, or fetal or newborn death within 6 weeks after birth; individual elements of the composite, the frequency of small for gestational age neonates, birthweight.
Neonatal healthcare utilization | 6 weeks
  NICU and hospital length of stay
Maternal morbidity | From randomization to 6 weeks after delivery, up to 20 weeks
  Composite of severe hypertension, pulmonary edema, heart failure, eclampsia, stroke, liver dysfunction, acute renal failure, thrombocytopenia, abruption, ICU admission, postpartum hospital readmission for hypertension management, or death within 6 weeks of delivery; individual elements of the composite.
Maternal healthcare utilization | From randomization to 6 weeks after delivery, up to 20 weeks
  Antepartum and postpartum hospital length of stay, ICU admission, postpartum readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sinkey, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Oschner, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stergiou GS, Alpert B, Mieke S, Asmar R, Atkins N, Eckert S, Frick G, Friedman B, Grassl T, Ichikawa T, Ioannidis JP, Lacy P, McManus R, Murray A, Myers M, Palatini P, Parati G, Quinn D, Sarkis J, Shennan A, Usuda T, Wang J, Wu CO, O'Brien E. A universal standard for the validation of blood pressure measuring devices: Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Collaboration Statement. J Hypertens. 2018 Mar;36(3):472-478. doi: 10.1097/HJH.0000000000001634. PMID 29384983
- [Background] Sinkey RG, Battarbee AN, Bello NA, Ives CW, Oparil S, Tita ATN. Prevention, Diagnosis, and Management of Hypertensive Disorders of Pregnancy: a Comparison of International Guidelines. Curr Hypertens Rep. 2020 Aug 27;22(9):66. doi: 10.1007/s11906-020-01082-w. PMID 32852691
- [Background] Ives CW, Sinkey R, Rajapreyar I, Tita ATN, Oparil S. Preeclampsia-Pathophysiology and Clinical Presentations: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Oct 6;76(14):1690-1702. doi: 10.1016/j.jacc.2020.08.014. PMID 33004135
- [Background] Battarbee AN, Sinkey RG, Harper LM, Oparil S, Tita ATN. Chronic hypertension in pregnancy. Am J Obstet Gynecol. 2020 Jun;222(6):532-541. doi: 10.1016/j.ajog.2019.11.1243. Epub 2019 Nov 9. PMID 31715148
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Bello NA, Woolley JJ, Cleary KL, Falzon L, Alpert BS, Oparil S, Cutter G, Wapner R, Muntner P, Tita AT, Shimbo D. Accuracy of Blood Pressure Measurement Devices in Pregnancy: A Systematic Review of Validation Studies. Hypertension. 2018 Feb;71(2):326-335. doi: 10.1161/HYPERTENSIONAHA.117.10295. Epub 2017 Dec 11. PMID 29229741
- [Background] Sinkey RG, Oparil S. Lower Blood Pressure Thresholds Raise the Bar in Pregnancy. Circ Res. 2019 Jul 5;125(2):195-197. doi: 10.1161/CIRCRESAHA.119.315384. Epub 2019 Jul 3. No abstract available. PMID 31268860
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Hauth JC, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Iams JD, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. First-trimester prediction of preeclampsia in nulliparous women at low risk. Obstet Gynecol. 2012 Jun;119(6):1234-42. doi: 10.1097/AOG.0b013e3182571669. PMID 22617589
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Hauth JC, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Grobman WA, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). The utility of uterine artery Doppler velocimetry in prediction of preeclampsia in a low-risk population. Obstet Gynecol. 2012 Oct;120(4):815-22. doi: 10.1097/AOG.0b013e31826af7fb. PMID 22996099
- [Background] Petersen EE, Davis NL, Goodman D, Cox S, Syverson C, Seed K, Shapiro-Mendoza C, Callaghan WM, Barfield W. Racial/Ethnic Disparities in Pregnancy-Related Deaths - United States, 2007-2016. MMWR Morb Mortal Wkly Rep. 2019 Sep 6;68(35):762-765. doi: 10.15585/mmwr.mm6835a3. PMID 31487273
- [Background] Tita AT, Szychowski JM, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson K, Haas DM, Plante L, Metz T, Casey B, Esplin S, Longo S, Hoffman M, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su E, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Geller NL, Oparil S, Cutter GR, Andrews WW; Chronic Hypertension and Pregnancy (CHAP) Trial Consortium. Treatment for Mild Chronic Hypertension during Pregnancy. N Engl J Med. 2022 May 12;386(19):1781-1792. doi: 10.1056/NEJMoa2201295. Epub 2022 Apr 2. PMID 35363951